CLINICAL TRIAL: NCT00427921
Title: A Multicentre, Open Label, Treatment Protocol of the Human Anti-TNF Monoclonal Antibody Adalimumab in Canadian Subjects With Moderate to Severe Crohn's Disease (ACCESS)
Brief Title: Human Anti-TNF Monoclonal Antibody Adalimumab in Canadian Subjects With Moderate to Severe Crohn's Disease (ACCESS)
Acronym: ACCESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Tom Koutsavlis, Medical Director, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W06-405
Record Dates: First submitted 2007-01-26; First posted 2007-01-29 (Estimated); Results first posted 2009-10-23 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Open Label
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — 160 mg loading dose, 80 mg at week 2, 40 mg every other week
  Other Names: ABT-D2E7; Humira

SUMMARY:
To make adalimumab available to subjects suffering from moderately to severely active Crohn's Disease (CD) and to expand the safety information on adalimumab. The study also assessed changes in Patient Reported Outcome Measures from baseline.

DETAILED DESCRIPTION:
This was a Phase 3, multicenter, open-label, Early Access Study with an induction regimen of adalimumab 160 mg subcutaneous (SC) at Baseline and 80 mg SC at Week 2, followed by maintenance dosing of 40 mg every other week (eow) starting at Week 4 in subjects with moderately to severely active Crohn's Disease (CD) who were eligible to receive biologic therapy or who had failed to respond to, lost response to, or were intolerant to infliximab. Failure of prior therapy was determined by the Investigator. Subjects were to have an 8-week wash-out period prior to Baseline from the last dose of infliximab.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years of age and older
* Females: Not of childbearing potential OR Practicing approved birth control throughout the study and for 150 days after study completion
* Diagnosis of moderate to severe CD for greater than 16 weeks prior to screening; Crohn's Disease Activity Index score > 220 OR Harvey Bradshaw Index equal to or higher than 7, and who are refractory to optimal conventional therapies such as, 5-aminosalicylic acid (5-ASA), glucocorticoids, and immunosuppressive therapies (azathioprine, 6-MP and MTX)
* Subjects who failed prior infliximab therapy (as determined by the primary investigator), including those who never clinically responded ("primary non-responders")

Exclusion Criteria:

* History of cancer other than some skin and cervical cancers
* History of opportunistic infections, central nervous system (CNS) demyelinating disease, chronic viral hepatitis, or untreated tuberculosis
* Subjects with other, poorly controlled medical conditions
* Subjects with any prior exposure to Tysabri® (natalizumab)
* Subjects who have received any investigational agent in the past 30 days or 5 half-lives prior to screening (whichever is longer)
* Female subjects who are pregnant or breast-feeding or considering becoming pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Baloukas, Study Director — Abbott; Remo Panaccione, MD, FRCPC, Study Chair — Director, Inflammatory Bowel Disease Clinic, Associate Professor of Medicine, University of Calgary, Calgary, AB, Canada
Locations (1):
- Global Medical Information - Abbott, Abbott Park, Illinois, United States

REFERENCES:
- See also: For more information, see attached website — http://www.humira.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- 40 mg Adalimumab Every Other Week: Induction regimen of adalimumab 160 mg subcutaneous (SC) at Baseline and 80 mg SC at Week 2, followed by maintenance dosing of 40 mg every other week (eow) starting at Week 4
Period: Overall Study
Arm/Group | 40 mg Adalimumab Every Other Week
Started | 304
Completed | 254
Not Completed | 50
Not completed — Adverse Event | 26
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 2
Not completed — Other reason not specified | 10
Not completed — Adverse Event + Hospitalization | 1
Not completed — Adverse Event + Withdrew Consent | 1
Not completed — Adverse Event + No Response | 1
Not completed — Adverse Event + Worsening of CD | 1
Not completed — Adverse Event + No Therapeutic Benefit | 1
Not completed — Adverse Event + Lost Response | 1
Not completed — Adverse Event + Withdrawn from Study | 1
Not completed — Withdrew Consent + Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | 40 mg Adalimumab Every Other Week
Number analyzed (Participants) | 304
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 296
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173
  Male | 131
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 291
  More than one race | 1
  Unknown or Not Reported | 6
  Hispanic | 0
Region of Enrollment [Number; unit: Participants]
  Canada | 304
Alcohol [Number; unit: participants]
  User | 147
  Ex-User | 15
  Non-User | 142
C-Reactive protein mg/dL [Number; unit: participants]
  < 1.0 mg/dL | 148
  > = 1.0 mg/dL | 155
  Missing | 1
Nicotine [Number; unit: participants]
  User | 98
  Ex-User | 84
  Non-User | 122
Number Subjects With Draining Cutaneous Fistulas at Screening [Number; unit: participants]
  Count 0 lesions | 235
  Count 1 lesion | 42
  Count 2 lesions | 16
  Count 3 lesions | 5
  Count >=4 lesions | 5
  Missing | 1
Number Subjects with Perianal Fistulas at Screening [Number; unit: Participants]
  Count 0 | 244
  Count 1 | 35
  Count 2 | 17
  Count 3 | 4
  Count >=4 | 3
  Missing | 1
Number of Subjects with Abdominal Fistulas at Screening [Number; unit: Participants]
  Count 0 | 291
  Count 1 | 10
  Count 2 | 1
  Count 3 | 0
  Count >=4 | 1
  Missing | 1
Summary of Locations of Crohn's Disease at Screening (All Treated Subjects) [Number; unit: participants] — Crohn's Disease may be at multiple locations
  participants
    Anal/Perianal | 2
    Colon | 40
    Gastroduodenum | 1
    Rectum | 3
    Jejunum | 2
    Ileum | 54
    Other | 3
    Ileum + Other | 7
    Jejunum + Ileum | 3
    Rectum + Ileum | 7
    Rectum + Ileum + Other | 1
    Gastroduodenum + Ileum | 3
    Colon + Other | 2
    Colon + Ileum | 64
    Colon + Ileum + Other | 3
    Colon + Jejunum + Ileum | 3
    Colon + Rectum | 8
    Colon + Rectum + Ileum | 13
    Colon + Rectum + Ileum + Other | 2
    Colon + Gastroduodenum + Ileum | 1
    Colon+GD+Jejunum+Ileum | 2
    Colon+GD+Rectum+ Other | 1
    Colon+GD+Rectum+Jejunum+Ileum | 1
    Anal/Perianal + Ileum | 16
    Anal/Perianal + Ileum + Other | 2
    Anal/Perianal + Jejunum + Ileum | 1
    Anal/Perianal + Rectum | 2
    Anal/Perianal + Rectum + Other | 1
    Anal/Perianal + Rectum + Ileum | 3
    Anal/Perianal + Colon | 6
    Anal/Perianal + Colon + Other | 2
    Anal/Perianal + Colon + Ileum | 13
    Anal/Perianal + Colon + Ileum + Other | 3
    Anal/Perianal + Colon + Jejunum + Ileum | 3
    Anal/Perianal + Colon + Rectum | 3
    Anal/Perianal + Colon + Rectum + Ileum | 13
    Anal/Perianal + Colon + Rectum + Ileum + Other | 2
    Anal/Perianal + Colon + Rectum +Jejunum + Ileum | 1
    Anal/Perianal + Colon + GD + Ileum | 4
    Anal/Perianal + Colon + GD +Rectum + Ileum | 2
    Anal/Perianal+Colon+GD+Rectum+Jejunum+Ileum | 1
Weight in kilograms [Number; unit: Participants]
  < = 70 kg | 163
  > 70 kg | 141
Duration of Crohn's Disease at Screening in Years [Mean (Standard Deviation); unit: years] | 11.8 (9.54)

OUTCOME MEASURES:

1. Primary Outcome: Mean Extent of Exposure - Duration in Days
Description: Extent of exposure for all adalimumab treated subjects
Time Frame: Up to 24 weeks
Population: In addition to the Intent To Treat population, summaries for outcome measures were provided for the analyzable subsets, and subjects in the Per-Protocol analysis set.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 40 mg Adalimumab Every Other Week
Number analyzed (Participants) | 304
days | 159.2 (34.78)

2. Post Hoc Outcome: Harvey-Bradshaw Index (HBI) Mean Change From Baseline
Description: HBI score (range 0-30) sum subtotal of 5 parameters of subject's CD activity: a)Well being 0=very well-4=terrible b) Abdominal pain 0=none- 3=severe c) Number liquid stools per day d) Abdominal mass 0=none-3=tender e) Complications: 1 point each. Decrease indicates improvement. Absolute decrease of 3 units on scale is clinically important.
Time Frame: Weeks 4, 8, 12, and 24, and Last Assessment Value (last nonmissing value)
Population: Intent to Treat - subjects who received at least one dose of study drug.
Measure: Mean (95% Confidence Interval); unit: Units on scale
Arm/Group | 40 mg Adalimumab Every Other Week
Number analyzed (Participants) | 304
Units on scale
  Week 4 | -4.39 [-4.94 to -3.84]
  Week 8 | -4.53 (5.175) [-5.12 to -3.93]
  Week 12 | -5.32 (5.008) [-5.90 to -4.74]
  Week 24 | -6.36 (5.031) [-6.96 to -5.75]
  Last Assessment Value | -5.92 (5.162) [-6.50 to -5.34]

3. Secondary Outcome: Fistula Count Mean Change From Baseline (Change in Number of Fistulas From Baseline).
Description: Draining fistula counts is the sum of abdominal and perianal fistulas for each subject at each visit.
Time Frame: Week 12, Week 24, and Last Assessment Value (last nonmissing value)
Measure: Mean (Standard Deviation); unit: number of fistulas
Arm/Group | 40 mg Adalimumab Every Other Week
Number analyzed (Participants) | 304
number of fistulas
  Week 12 | -0.17 (0.644)
  Week 24 | -0.15 (0.587)
  Last Assessment Value | -0.15 (0.567)

4. Primary Outcome: Total Number of Injections of Adalimumab
Description: Extent of exposure for all adalimumab treated subjects
Time Frame: Up to 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: injections
Arm/Group | 40 mg Adalimumab Every Other Week
Number analyzed (Participants) | 304
injections
  Number of Injections During Induction Therapy | 2 (0.1)
  Number of Injections During Maintenance Therapy | 11.8 (4.24)

5. Primary Outcome: Compliance With Number of Injections of Adalimumab. Compliance Corresponds to Patients Who Received Their Injections.
Description: Treatment compliance (%) = 100 * (Number of doses of study medication actually received)/(Number of doses planned during the subject's participation in the study).
Time Frame: Up to 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of injections
Arm/Group | 40 mg Adalimumab Every Other Week
Number analyzed (Participants) | 304
Percentage of injections | 98.85 (4.207)

6. Post Hoc Outcome: Short Inflammatory Bowel Disease Questionnaire (SIBDQ) Mean Change From Baseline
Description: Quality of life questionnaire for patients with IBD consisting of 4 domains: systemic, social, emotional, and bowel. This is a 10-item questionnaire, and all items are reported with a 7-point scale (ranging from 1 = poor HRQOL, to 7 = optimum HRQOL). Total SIBDQ score ranges from 10 (quality of life has been negatively affected tremendously by IBD) to 70 (quality of life is barely impacted by IBD). A change greater than 9 points was the minimal clinically important difference (MCID).
Time Frame: Weeks 4, 8, 12, and 24, and Last Assessment Value (last nonmissing value)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 40 mg Adalimumab Every Other Week
Number analyzed (Participants) | 304
units on a scale
  Week 4 | 10.16 (10.692)
  Week 8 | 11.85 (11.591)
  Week 12 | 13.14 (11.783)
  Week 24 | 15.06 (12.209)
  Last Assessment Value | 13.74 (12.629)

7. Secondary Outcome: Overall Health Care Resource Utilization
Description: From the "Overall Health Care Resource Utilization Questionnaire": Number visits to physician, number visits to Emergency Room, number of hospital admissions, number of days of hospitalization.
Time Frame: Up to 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | 40 mg Adalimumab Every Other Week
Number analyzed (Participants) | 304
number of visits
  Number of visits to a physician | 1.13 (2.794)
  Number of visits to Emergency Room | 0.17 (0.522)
  Number of hospital admissions | 0.10 (0.346)
  Number of days of hospitalizations | 0.60 (2.790)

8. Secondary Outcome: Employment Status: Number of Subjects Employed
Description: Summary of employment status of those employed.
Time Frame: Baseline, Weeks 4, 8, 12, and 24, and Last Assessment Value (last nonmissing value)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 40 mg Adalimumab Every Other Week
Number analyzed (Participants) | 304
participants
  Baseline | 195 (64.1)
  Week 4 | 199
  Week 8 | 198
  Week 12 | 192
  Week 24 | 190
  Last Assessment Value | 208

9. Secondary Outcome: 50% Improvement in Draining Fistula Count and Fistula Healing
Description: Decrease in draining fistula is beneficial. "50 percent improvement" refers to a reduction in the number of baseline fistula by 50 percent.
Time Frame: Week 12, Week 24, Last Assessment Value (last nonmissing value)
Population: Intent To Treat
Measure: Number; unit: participants
Arm/Group | 40 mg Adalimumab Every Other Week
Number analyzed (Participants) | 62
participants
  Week 12 50% Improvement in draining fistula | 35
  Week 24 50% Improvement in draining fistula | 31
  Last Value 50% Improvement in draining fistula | 32
  Week 12 Fistula Healing | 23
  Week 24 Fistula Healing | 27
  Last Assessment Value Fistula Healing | 28

10. Secondary Outcome: Work Productivity and Activity Impairment - Change From Baseline in Overall Work Impairment
Description: Scores are expressed as impairment percentages, higher numbers indicate greater impairment and less productivity (0% = no impairment; 100% = total loss of work productivity).
  Minimal clinically important difference = 7 points. Measure is Mean percent change.
Time Frame: Weeks 4, 8, 12, and 24, and Last Assessment Value (last nonmissing value)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | 40 mg Adalimumab Every Other Week
Number analyzed (Participants) | 304
Units on scale
  Week 4 | -22.08 (28.454)
  Week 8 | -22.36 (29.337)
  Week 12 | -29.93 (33.669)
  Week 24 | -31.23 (30.403)
  Last Assessment Value | -28.49 (32.286)

11. Secondary Outcome: Hematology - Change From Baseline to Final Visit
Description: Changes from the Group mean at baseline are compared to the final visit Group mean value
Time Frame: Up to 24 weeks
Measure: Mean (Standard Deviation); unit: number
Arm/Group | 40 mg Adalimumab Every Other Week
Number analyzed (Participants) | 304
number
  Hemoglobin (g/L) | 2.2 (12.43)
  Hematocrit (fraction) | 0.011 (0.0376)
  Red blood cell count (x10^9/L) | 0.03 (0.353)
  Platelet Count (x10^9/L) | -30.2 (89.28)
  White blood cell count (x10^9/L) | -1.59 (3.297)
  Neutrophils (x10^9/L) | -2.005 (3.1777)
  Lymphocytes (x10^9/L) | 0.408 (0.7285)
  Monocytes (x10^9/L) | -0.014 (0.1725)
  Eosinophils (x10^9/L) | 0.009 (0.1505)
  Basophils (x10^9/L) | -0.015 (0.0617)

12. Secondary Outcome: Clinical Chemistry - Change From Baseline to Final Visit
Description: Changes from the Group mean at Baseline are compared to the final visit Group mean value
Time Frame: Up to 24 weeks
Measure: Mean (Standard Deviation); unit: number
Arm/Group | 40 mg Adalimumab Every Other Week
Number analyzed (Participants) | 304
number
  SGPT/ALT (U/L) | 0.6 (17.89)
  SGOT/ALT (U/L) | 1.6 (10.35)
  Alkaline phosphatase (U/L) | -5.2 (21.53)
  Total Bilirubin (mcmol/L) | 1.6 (4.06)
  Creatinine (mcmol/L) | 1.7 (10.35)
  BUN (mmol/L) | 0.06 (1.367)
  Uric acid (mcmol/L) | 4.6 (52.38)
  Inorganic phosphate | 0.016 (0.2588)
  Calcium (mmol/L) | 0.008 (0.1189)
  Sodium (mmol/L) | -0.3 (2.38)
  Potassium (mmol/L) | -0.00 (0.779)
  Albumin (G/L) | 0.4 (4.01)
  Total protein (G/L) | 0.8 (4.83)
  Cholesterol (mmol/L) | 0.021 (0.7024)
  Triglycerides (mmol/L) | 0.093 (0.7581)
  C-reactive protein (mg/L) | -8.181 (28.7023)
  Glucose - fasting (mmol/L) | -0.268 (1.3893)

13. Secondary Outcome: Urinalysis - Change From Baseline to Final Visit
Description: Changes from the Group mean at baseline are compared to the final visit Group mean value
Time Frame: Up to 24 weeks
Measure: Mean (Standard Deviation); unit: number
Arm/Group | 40 mg Adalimumab Every Other Week
Number analyzed (Participants) | 304
number
  Urine pH | 0.02 (0.980)
  Specific gravity | -0.0004 (0.00713)

14. Secondary Outcome: Work Productivity and Activity Impairment - Change From Baseline in Absenteeism
Description: The Work Productivity and Activity Impairment (WPAI) questionnaire is a validated, self-administered tool used to assess the impact of disease on productivity. There are four component scores for WPAI: absenteeism, presenteeism, total work productivity impairment, daily activity impairment. The score for each component ranges from 0% to 100% (0%=no impairment; 100%=total loss of work productivity or activity). The minimal clinically important difference (MCID) is an absolute change of 7%.
Time Frame: Weeks 4, 8, 12, and 24, and Last Assessmentl Value (last nonmissing value)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 40 mg Adalimumab Every Other Week
Number analyzed (Participants) | 304
units on a scale
  Week 4 | -5.99 (24.592)
  Week 8 | -7.55 (27.543)
  Week 12 | -8.74 (33.477)
  Week 24 | -8.54 (27.260)
  Last Assessment Value | -6.46 (29.167)

15. Secondary Outcome: Work Productivity and Activity Impairment - Change From Baseline in Presenteeism
Description: as for outcome 14
Time Frame: Weeks 4, 8, 12, and 24, and Last Assessment Value (last nonmissing value)
Population: In addition to the ITT population, summaries for outcome measures were provided for the analyzable subsets, and subjects in the Per-Protocol analysis set.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | 40 mg Adalimumab Every Other Week
Number analyzed (Participants) | 304
Units on scale
  Week 4 | -20.58 (26.115)
  Week 8 | -19.94 (27.151)
  Week 12 | -25.79 (30.113)
  Week 24 | -28.96 (28.472)
  Last Assessment Value | -26.69 (30.058)

16. Secondary Outcome: Work Productivity and Activity Impairment - Change From Baseline in Activity Impairment
Description: as for outcome 14
Time Frame: Weeks 4, 8, 12, and 24, and Last Assessment Value (last nonmissing value)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | 40 mg Adalimumab Every Other Week
Number analyzed (Participants) | 304
Units on scale
  Week 4 | -23.59 (26.928)
  Week 8 | -24.79 (28.431)
  Week 12 | -30.36 (28.697)
  Week 24 | -34.00 (29.552)
  Last Assessment Value | -30.98 (30.484)

ADVERSE EVENTS:
Arm/Group | 40 mg Adalimumab Every Other Week
Serious Adverse Events (participants affected / at risk) | 44
Other Adverse Events (participants affected / at risk) | 133
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | 40 mg Adalimumab Every Other Week
anaemia (Blood and lymphatic system disorders) | 3/304
heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1/304
atroventricular block complete (Cardiac disorders) | 1/304
abdominal pain (Gastrointestinal disorders) | 2/304
Crohn's Disease (Gastrointestinal disorders) | 13/304
GI haemorrhage (Gastrointestinal disorders) | 1/304
GI motility disorder (Gastrointestinal disorders) | 1/304
ileal perforation (Gastrointestinal disorders) | 1/304
internal hernia (Gastrointestinal disorders) | 1/304
small intestinal obstruction (Gastrointestinal disorders) | 9/304
subileus (Gastrointestinal disorders) | 2/304
death (General disorders) | 1/304
fatigue (General disorders) | 1/304
inflammation (General disorders) | 1/304
abdominal abscess (Infections and infestations) | 4/304
appendicitis (Infections and infestations) | 1/304
perianal abscess (Infections and infestations) | 1/304
pneumonia legionella (Infections and infestations) | 1/304
rectal abscess (Infections and infestations) | 1/304
anastomotic complication (Injury, poisoning and procedural complications) | 1/304
anatomotic leak (Infections and infestations) | 1/304
anastomotic stenosis (Injury, poisoning and procedural complications) | 1/304
haemoglobin decreased (Investigations) | 1/304
intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1/304
fistula (Musculoskeletal and connective tissue disorders) | 1/304
lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/304
anxiety (Psychiatric disorders) | 1/304
nephrolithiasis (Renal and urinary disorders) | 1/304
renal colic (Renal and urinary disorders) | 1/304
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/304
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1/304
pulmonary emolism (Respiratory, thoracic and mediastinal disorders) | 1/304
dyshidrosis (Skin and subcutaneous tissue disorders) | 1/304
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | 40 mg Adalimumab Every Other Week
Abdominal pain (Gastrointestinal disorders) | 23/304
Nausea (Gastrointestinal disorders) | 19/304
Headache (Nervous system disorders) | 19/304
Arthralgia (Musculoskeletal and connective tissue disorders) | 18/304
Nasopharyngitis (Infections and infestations) | 15/304
Fatigue (General disorders) | 14/304
Injection site reaction (General disorders) | 23/304
Crohn's Disease (Gastrointestinal disorders) | 49/304

LIMITATIONS AND CAVEATS:
Subjects who failed prior infliximab therapy were eligible to enter study after minimum 8 week wash-out since last dose. Includes subjects who previously used infliximab & never responded or responded & developed intolerance/lost efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Responsibility of preparation and maintenance of the single database, first publication, and, presentation of Study shall reside with Abbott. No independent manuscript may be submitted for publication until first manuscript has been accepted for publication or twelve (12) months after completion of the Study at all sites, which ever occurs first.